CLINICAL TRIAL: NCT01381276
Title: Vitamin A Equivalence of Carotenoids From Cassava in Women
Brief Title: Vitamin A Absorption From Cassava in Women
Acronym: FL-80
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: USDA, Western Human Nutrition Research Center (U.S. Federal Agency)
Collaborators: HarvestPlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: WHNRC 223773-1
Record Dates: First submitted 2011-06-22; First posted 2011-06-27 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2011-12

CONDITIONS: Vitamin A Deficiency
Keywords: Vitamin A
MeSH Terms: conditions — Vitamin A Deficiency | interventions — Oils

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cassava Treatment 1 (Experimental): Single meal containing bio-fortified, high carotenoid cassava without oil.
  Interventions: Other: Beta-Carotene bio-fortified cassava porridge without oil
- Cassava Treatment 2 (Experimental): Single meal containing bio-fortified, high carotenoid cassava with oil.
  Interventions: Other: Beta-Carotene bio-fortified cassava porridge with oil
- Cassava Treatment 3 (Active Comparator): Single meal containing low carotenoid cassava with oil and retinyl palmitate.
  Interventions: Other: White cassava porridge with retinyl palmitate reference dose

INTERVENTIONS:
Other: Beta-Carotene bio-fortified cassava porridge without oil — 300 g of porridge (11 ounces) containing 100 g drained mashed cassava and approximately 1 mg beta-carotene.
  Arms: Cassava Treatment 1
Other: Beta-Carotene bio-fortified cassava porridge with oil — 300g porridge (11 ounces) containing 100 g drained mashed cassava, 15 g peanut oil, and approximately 1 mg beta-carotene.
  Arms: Cassava Treatment 2
Other: White cassava porridge with retinyl palmitate reference dose — 300 g porridge containing 15 mL peanut oil, 100 g drained mashed cassava, and a tracer of approximately .3 mg pure food-grade retinyl palmitate.
  Arms: Cassava Treatment 3

SUMMARY:
The purpose of this study is to determine the vitamin A equivalents in high-carotenoid varieties of cassava.

DETAILED DESCRIPTION:
We plan to conduct a single site intervention phase II intervention study in healthy adult women. Women will serve as their own controls, and will be fed three treatments in random order: a single meal of low-carotenoid cassava porridge with fat, a similar meal of bio-fortified cassava (that is high in vitamin A-forming carotenoids) with fat, and a similar meal of bio-fortified cassava without fat. Carotenoids and vitamin A will be measured in the triacylglycerol-rich lipoprotein (TRL) fraction of plasma by standard methods involving ultracentrifugation (to concentrate the TRL fraction) followed by reversed-phase HPLC using electrochemical detection. We plan to collect sufficient data to identify the times of the first appearance and peak concentrations in retinol, retinyl esters, alpha-carotene (AC), beta-carotene (BC), beta-carotene isomers (BCI), and cryptoxanthin (CX) in TRL: when a single meal containing moderately high amounts of carotenoids from bio-fortified cassava is fed to healthy adult women. We will use this data to determine the vitamin A equivalency of bio-fortified cassava in adult women, and the effect of fat on vitamin A equivalency of bio-fortified cassava.

ELIGIBILITY:
Inclusion Criteria:

* non-smoking
* BMI between 18-30
* total cholesterol concentrations between 90 and 225 mg/dL
* blood pressure under 140/90 mm Hg
* hemoglobin above 11.5 g/dL
* blood chemistries within the normal range

Exclusion Criteria:

* must not be pregnant or trying to get pregnant
* must not be taking fat, triacylglycerol, or cholesterol lowering medications) such as orlistat, gemfibrozil, niacin, lovastatin, simvastatin, colestipol, and ezetimibe)
* must not taking medicines containing high doses of retinoids such as Accutane or high vitamin A or carotenoid supplements
* must not have blood chemistry or health history results consistent with acute cancer or heart disease
* no obvious psychological or sociological problems such as alcoholism, drug abuse, or severe and acute mental illness that would influence their ability to sign an informed consent agreement or to participate in study duties and activities
* must not be allergic to cassava, peanuts, or peanut oil

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Vitamin A equivalency from varieties of cassava with and without oil | 0, 60, 150, 240, 330, 420, 510, 600, 1440 min
  Vitamin A and other carotenoids will be measured in triacylglycerol rich lipoprotein fractions at 0, 60, 150, 240, 330, 420, 510, 600, and 1440 minutes after consumption of cassava containing meal.

CONTACTS AND LOCATIONS:
Overall Officials: Betty J Burri, PhD, Principal Investigator — WHNRC, ARS, University of California Davis
Locations (1):
- Western Human Nutrition Center, University of California Davis, Davis, California, United States